CLINICAL TRIAL: NCT05176535
Title: Study to Determine Vaginal Colonization and Effect of an Oral Probiotic That Contains L.Rhamnosus, L. Plantarum and L. Crispatus in Women (PROSALVAG)
Brief Title: Determination of Vaginal Colonization and the Effect of an Oral Probiotic (PROSALVAG)
Acronym: PROSALVAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertypharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-FBB-07
Record Dates: First submitted 2021-11-30; First posted 2022-01-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-07

CONDITIONS: Microbial Colonization; Dysbiosis; Fertility Issues
MeSH Terms: conditions — Communicable Diseases; Dysbiosis; Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FertyBiotic Balance (Experimental): Participants received FertyBiotic Balance one capsule a day
  Interventions: Dietary Supplement: FertyBiotic Balance

INTERVENTIONS:
Dietary Supplement: FertyBiotic Balance — Lactobacillus rhamnosus BPL 205, Lactobacillus plantarum BPL207 and Lactobacillus crispatus BPL209

SUMMARY:
The aim of this study is to determine the efficacy of an oral nutraceutical with probiotics in restore vaginal health.

DETAILED DESCRIPTION:
After being informed about the study, all patients meeting the inclusion/exclusion criteria and giving written informed consent will receive a nutraceutical containing L. rhamnosus, L. plantarum and L. crispatus once daily.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 35-43 years old
* Vaginal pH > 4,5 and low Lactobacillus count or Nugent score of 4-6
* With interest in getting pregnant and ideally in IVF waiting list
* History of recurrent genitourinary infections

Exclusion Criteria:

* Any pathology that interferes with the study
* Current intake of food supplements or probiotics
* Current intake of contraceptives
* Use of oral or vaginal probiotics in the last 6 months
* Hypersensitivity to any of the components of the studied product
* Current vaginal infection
* Pregnant women
* Breastfeeding
* Use of intrauterine device
* Use of spermicide
* Use of cervical caps as hormonal therapy

Ages: 35 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Restoration of vaginal microbiota
Enrollment: 32 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Rectal and vaginal colonization | 10 weeks
  Rectal and vaginal colonization will be evaluated by measuring massive sequencing of 16SrRNA gen

SECONDARY OUTCOMES:
Autoinmune capacity | 10 weeks
  Autoinmune capacity will be evaluated by measuring plasma levels of IL-10, TNF- alpha and IL-10
Antioxidant effect | 10 weeks
  Antioxidant will be evaluated by measuring Total Antioxidant Capacity (TAC) and Malondialdehyde

CONTACTS AND LOCATIONS:
Locations (1):
- HM Fertility Centter Vallés, Alcalá de Henares, Madrid, Spain